CLINICAL TRIAL: NCT00138775
Title: D-Serine Adjuvant Pharmacotherapy for the Treatment of Schizophrenia
Brief Title: Israel Multicenter D-Serine Study (IMSER) for the Treatment of Schizophrenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-03-3093-MW-CTIL
Record Dates: First submitted 2005-08-28; First posted 2005-08-30 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: D-serine; Negative symptoms; Cognition; Schizophrenia; Amino acid
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Drug: D-serine

SUMMARY:
The goal of the present study is to evaluate the effect of D-serine, added to antipsychotic treatment, on negative and cognitive symptoms in schizophrenia.

The investigators are hypothesizing that D-serine will improve cognitive functioning and negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV) diagnosis of schizophrenia and\or schizoaffective disorder.
* Age between 18 to 64.
* PANSS negative symptom score higher than 19.
* SAS total score lower than 12.
* CDSS suicidal risk lower than 2

Exclusion Criteria:

* Epilepsy
* Meets DSM-IV criteria for mental retardation.
* Medical condition which confounds presentation or treatment (e.g. uncontrolled diabetes mellitus, history of kidney stones, acute drug toxicity, dementia, delirium, stroke, etc.)
* Meets DSM-IV criteria for alcohol or drug dependence in last 6 months.
* Meets DSM-IV criteria for alcohol or drug abuse in last one month.
* Treatment with clozapine.
* Current positive pregnancy test or not using acceptable method of birth control.
* Meets DSM-IV criteria for current anxiety or mood disorders

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2004-10; Study Completion 2007-10

PRIMARY OUTCOMES:
SANS - Scale for the Assessment of Negative Symptoms - weeks 0, 8 and 16
Measurement and Treatment Research for Cognition in Schizophrenia (MATRICS) battery - visit weeks 0, 8 and 16

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale of Schizophrenia (PANSS) positive, negative, general and total score - weeks 0, 8 and 16
Simpson-Angus Scale (SAS) total score - weeks 0, 8 and 16
Clinical Global Impressions (CGI) score - weeks 0, 8 and 16
Calgary Depression Scale for Schizophrenia (CDSS) score - weeks 0, 8 and 16
Side effect check list

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, MD, Principal Investigator — Sheba Medical Center
Locations (14):
- Israel (14):
  - Mazra Mental Health Center, Acre
  - Ha-Emek Medical Center, Afula
  - Abarbanel Mental Health Center, Bat Yam
  - Beer-Yaacov Mental Health Center, Beer-Yaacov
  - Shalvata Mental Health Center, Hod HaSharon
  - Kfar Shaul Psychiatric Hospital, Jerusalem
  - The Sarah Herzog Memorial Hospital, Jerusalem
  - Nes-Ziona Mental Health Center, Ness Ziona
  - Lev Hasharon Mental Health Center, Pardesiyya
  - Geha Mental Health Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Shaar Menashe Mental Health Center, Shaar Menashe
  - Jaffa Mental Health Center, Tel Aviv
  - Maccabi Mental Health Center, Tel Aviv

REFERENCES:
- [Derived] Weiser M, Heresco-Levy U, Davidson M, Javitt DC, Werbeloff N, Gershon AA, Abramovich Y, Amital D, Doron A, Konas S, Levkovitz Y, Liba D, Teitelbaum A, Mashiach M, Zimmerman Y. A multicenter, add-on randomized controlled trial of low-dose d-serine for negative and cognitive symptoms of schizophrenia. J Clin Psychiatry. 2012 Jun;73(6):e728-34. doi: 10.4088/JCP.11m07031. PMID 22795211